CLINICAL TRIAL: NCT05713240
Title: REgiStry in Chinese yoUng pEople With Sudden Cardiac Death（RESCUE-SCD）
Brief Title: REgiStry in Chinese yoUng pEople With Sudden Cardiac Death
Acronym: RESCUE-SCD
Status: Not yet recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lei.Song,MD.&ph.D, Principal Investigator, Clinical Professor, China National Center for Cardiovascular Diseases
Other Study IDs: RESCUE-SCD
Record Dates: First submitted 2023-01-13; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Sudden Cardiac Death
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The number of sudden cardiac death is up to 540,000 every year in China. Inherited cardiovascular disease is a common cause of sudden cardiac death in young people, and diseases often have the characteristics of family aggregation, so it has a huge psychological and economic burden on family members. Studying the etiology of sudden cardiac death from the molecular level under the model of precision medicine is helpful for screening patients and their relatives so as to further diagnosis, treatment and management, which has important clinical and social significance.

DETAILED DESCRIPTION:
In this study, sudden cardiac death and high risk of sudden cardiac death in patients younger than 40 years of age are recruited prospectively after informed consent was given. The investigator will collect the baseline clinical characteristics of the patients at enrollment, including comprehensive physical examination, laboratory testing of blood and urine, electrocardiography, 24-hour Holter, echocardiography, MRI and other examinations if necessary. The specimens retained include blood or oral swabs for all patients, and myocardium for patients receiving autopsy. Genetic testing will be performed to identify carried disease genes, genetic risk factors and potential therapy targets.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sudden cardiac death and sudden unexplained death diagnosed according current practice guidelines.
* Patients at high risk for sudden cardiac death. (1) Family history of sudden cardiac death at a young age; （2）Successful resuscitation from cardiac arrest; （3) Implantable cardioverter defibrillator implantation after a comprehensive clinical assessment of high risk of sudden cardiac death.

Exclusion Criteria:

* Patients who refuse to sign the informed consent or decline follow-up.
* Patients with sudden death due to car accidents, electric shocks, drowning, fighting, carbon monoxide poisoning and other external causes.
* Patients with sudden death due to other definite causes, such as cerebrovascular accident, severe kidney disease, respiratory disease, neurological disease, etc.

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Sudden cardiac death and high risk of sudden cardiac death in patients younger than 40 years of age from multiple centers in China between March 1, 2023 and March 1, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
number of participants with cardiovascular deaths | an average of 2 years
  including sudden cardiac death and deaths due to heart failure and stroke

SECONDARY OUTCOMES:
number of participants with heart failure | an average of 2 years
  progress to level III or IV in New York Heart Association class
number of participants with stroke | an average of 2 years
  including cerebral infraction and hemorrhage
number of participants with myocardial infarction | an average of 2 years
  including ST-segment elevation myocardial infarction and non-ST-segment elevation myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided